CLINICAL TRIAL: NCT06800157
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled Phase IIa Study to Evaluate the Efficacy, Safety, and Tolerability of LW402 Tablets in Patients With Moderate to Severe Active Rheumatoid Arthritis
Brief Title: Study of LW402 Tablets in Moderate to Severe Rheumatoid Arthritis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Longwood Biopharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LW402-II-01
Record Dates: First submitted 2024-10-11; First posted 2025-01-29 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-01

CONDITIONS: Arthritis, Rheumatoid
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- LW402 50 mg (Experimental): LW402 50mg BID, combined with MTX
  Interventions: Drug: Drug: LW402; Drug: MTX
- Drug: LW402 125mg (Experimental): LW402 125mg BID, combined with MTX
  Interventions: Drug: Drug: LW402; Drug: MTX
- Placebo (Placebo Comparator): LW402 placebo BID, combined with MTX
  Interventions: Drug: Other: placebo; Drug: MTX

INTERVENTIONS:
Drug: Drug: LW402 — Oral tablets administered BID
  Arms: Drug: LW402 125mg; LW402 50 mg
Drug: Other: placebo — Placebo to match LW402 administered BID
  Arms: Placebo
Drug: MTX — Background treatment with MTX once a week

SUMMARY:
This Phase IIa study is designed to evaluate the dose-response relationship, efficacy, safety, and tolerability of LW402 tablets administered for 12 weeks in adult patients with active rheumatoid arthritis receiving background methotrexate (MTX) therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent;
2. The patient voluntarily accept and is able to follow the protocol procedures including medication and follow-up examination;
3. Age from 18 to 65 years old (including critical value), male or female;
4. Have a diagnosis of adult-onset rheumatoid arthritis (RA) as defined by American College of Rheumatology/ European League Against Rheumatism (ACR/EULAR) 2010 criteria for the classification of RA;
5. Diagnosisof moderately to severely active rheumatoid arthritis who also meets the following disease activity criteria at screening:

   * 6 swollen joints (based on 66 joint counts) and ≥ 6 tender joints (based on 68 joint counts) ;C-Reactive Protein (CRP) ≥ 10 mg/L or Eerythrocyte sedimentation rate（ESR）≥ 28 mm/h; DAS28-CRP>3.2；
6. Subjects had been on methotrexate (MTX) for ≥12 weeks and on a stable oral dose (7.5-25 mg/ week) of MTX for ≥4 weeks prior to randomization and are able to continue a stable dose of MTX during the study.

Exclusion Criteria:

1. Suspected or confirmed allergy to investigational drugs (including excipient and similar drugs) ,and other serious allergic diseases (except RA) judged by the investigator that may impair the safety of the subjects;
2. Had any inflammatory joint disease or autoimmune disease other than RA at screening (such as Gout, Reactive arthritis, Psoriatic arthritis, Spinal arthritis, Systemic lupus erythematosus, Mixed connective tissue diseases, etc.);
3. Have a history of lymphoproliferative disease; or have a current malignancy or history of malignancy (except Cutaneous squamous cell carcinoma in situ, Basal cell carcinoma or cervical carcinoma in situ, which have not shown any signs of recurrence for more than 5 years after achieving complete remission following radical treatment);
4. Have a history of major organ transplant (e.g., heart, lung, kidney, liver) or hematopoietic stem cell or bone marrow transplant;
5. Patients with Active tuberculosis at screening should be excluded.After a minimum of 4 weeks of treatment with 0.3g qd of isoniazid(or other prophylactic anti-tuberculosis treatments) for latent tuberculosis infection, continued screening could be considered when the investigator reassessed that the risk was controlled;
6. Presence of active infection, or have a history of: Systemic anti-infective treatment within 4 weeks prior to randomization; Sore throat, nasal congestion, acute upper respiratory tract infection, or systemic acute infection within 2 weeks prior to randomization; Presence of recurrent, chronic or other active infections in the screening period which may increase the risk of the subjects according to the evaluation of the investigators;
7. Have a history of recurrent herpes zoster, disseminated herpes zoster, or disseminated herpes simplex, or have a history of herpes zoster or herpes simplex within 2 months before randomization;
8. Presence of other diseases at screening that may interfere with the study evaluation;
9. Abnormal laboratory values at screening:

   Hemoglobin <10.0g/dL（100.0g/L） for male or < 9.0g/dL (90.0g/L) for female;WBC count <3.0×109/L;Neutrophil count <1.5×109/L; Platelet count <100×109/L; Lymphocyte count <0.5×109/L; Alanine transaminase (ALT) and/or Serum aspartate transaminase (AST) >1.5 upper limit of normal (ULN); Serum creatinine >1.5×upper limit of normal (ULN).
10. Positive for hepatitis B surface antigen and/or positive for hepatitis B core antibody (except HBV DNA negative or less than 500IU/ml) , positive for hepatitis C virus (HCV) antibody, positive for anti-human immunodeficiency virus (HIV) antibody, or anti-syphilis spiral antibody (except for TP-Ab positive but RPR or TRUST negative) at screening；
11. Have screening electrocardiogram (ECG) abnormalities that, in the opinion of the investigator , are clinically significant and indicate an unacceptable risk for the participant's participation in the study;
12. Previous use of any of the following medications or treatments:

    1. Have received potent opioids within 1 week before randomization;
    2. Have received any JAK inhibitor within 2 weeks before randomization;
    3. Have received any drugs that may interact with this product within 4 weeks before randomization, such as potent inhibitors of CYP3A4 (such as ketoconazole, itraconazole, clarithromycin, nefazodone, telithromycin, etc.), potent inducers of CYP3A4 (such as rifampicin);
    4. Have received disease-modifying antirheumatic drugs (DMARDs) or biological agents other than MTX. before randomization:

       Have received sulfasalazine, antimalarial drugs, penicillamine, oral gold salts, cyclosporine, azathioprine, cyclophosphamide, iguratimod, etc., within 4 weeks before randomization or no more than 5 half-life periods; Have received herbal medicines (including tripterygium wilfordii preparations, total glucosides of paeony, sinomenine and/or Chinese herbs) within 4 weeks before randomization; Have received Flunomide within 8 weeks before randomization; Have received TNF-α inhibitor (fusion protein) within 4 weeks, or received TNF-α inhibitor (monoclonal antibody) or abatacept within 12 weeks prior to randomization have received Tocilizumab within 10 weeks prior to randomization; Have received Rituximab within 24 weeks, or received another biologic agent with no more than 5 half-life periods before randomization.
    5. Are currently receiving receiving non-steroidal anti-inflammatory drugs (NSAIDs) before randomization with an unstable dosing regimen within 4 weeks before randomization;
    6. Are currently receiving corticosteroids at doses >10 mg per day of prednisone (or equivalent) or have been receiving an unstable dosing regimen of corticosteroids t within 4 weeks before randomization;
    7. Has been treated with intra-articular, intramuscular, intravenous, trigger point or tender point, intra-bursa, or intra-tendon sheath corticosteroids in the preceding 4 weeks prior to randomization;
13. Have been enrolled in another clinical study within 4 weeks or been treated by the last dose of any investigational drug within 5 half-lives prior to randomization;
14. Have been exposed to a live/attenuated vaccine within 8 weeks prior to randomization or are expected to need/receive a live/attenuated vaccine during the course of the study;
15. Have a history of drug or alcohol abuse (defined as consuming more than 28 units of alcohol per week. 1 unit =285ml beer or 25ml spirits containing at least 40% alcohol or 1 glass of wine) within the last 6 months.
16. Have donated ≥300mL of blood within 4 weeks prior to screening (except physiological blood loss in female) or plan to donate blood during or within 4 weeks after the study;
17. Women and/or men of childbearing potential and their partners who refuse to use effective contraception from the time they sign the informed consent until 6 months after the last dose, or who are planning to have children, donate eggs (women) or donate sperm (men);
18. Female who is pregnant or breastfeeding;
19. Other situations which are not suitable for the study per Investigator judgment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2023-02-27 (Actual); Primary Completion 2024-05-26 (Actual); Study Completion 2024-08-30 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in DAS28-CRP at Week 12 | 12 Weeks
  The DAS28-CRP is a composite measure of rheumatoid arthritis disease activity ranging from 0.0 to 9.4, calculated using tender joint count (28 joints), swollen joint count (28 joints), Patient's Global Assessment of Disease Activity (0-100 mm), and C-reactive protein (mg/L). Higher scores indicate greater disease activity.

SECONDARY OUTCOMES:
Proportion of patients achieving ACR20 response at Week 12 | 12 Weeks
  ACR20 is defined as at least 20% improvement in tender and swollen joint counts and improvement in at least 3 of 5 additional core measures (Patient Global Assessment, Physician Global Assessment, Pain, Disability/HAQ, and CRP)
Proportion of patients achieving ACR50 response at Week 12 | 12 Weeks
  ACR50 is defined as at least 50% improvement in tender and swollen joint counts and improvement in at least 3 of 5 additional core measures.
Proportion of patients achieving ACR70 response at Week 12 | 12 Weeks
  ACR70 is defined as at least 70% improvement in tender and swollen joint counts and improvement in at least 3 of 5 additional core measures.
Change from baseline in Health Assessment Questionnaire-Disability Index (HAQ-DI) at Week 12 | 12 Weeks
  HAQ-DI assesses physical function in patients with rheumatoid arthritis. HAQ-DI has a score range from 0-3. Higher scores indicate greater disability.
Incidence of treatment-emergent adverse events (TEAEs) | 16 Weeks
  All adverse events occurring after the first dose of study drug are recorded and summarized.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China